CLINICAL TRIAL: NCT00727129
Title: Placebo-Controlled, Randomized, Double-Blind, Multicenter Study, to Demonstrate the Efficacy of 12 Weeks of Treatment With USL-221 on Moderate to Severe Vasomotor Symptoms and Vulvar/Vaginal Atrophy in Postmenopausal Patients
Brief Title: Study to Evaluate Divigel for the Treatment of Postmenoupausal Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Upsher-Smith Laboratories (Industry)
Responsible Party: Upsher-Smith (Medical Affairs), Upsher-Smith Laboratories
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04-001
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Postmenopausal Symptoms
Keywords: vasomotor symptoms; estrogen; estradiol; hot flashes
MeSH Terms: conditions — Hot Flashes | interventions — Estradiol

INTERVENTIONS:
Drug: Divigel

SUMMARY:
The purpose of this study is to compare the safety and efficacy of USL-221 to placebo for postmenopausal patients.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Have moderate to severe hot flashes
* Normal Pap Smear

Exclusion Criteria:

* Abnormal mammogram
* Abnormal clinical breast exam
* BMI >35

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2004-07; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Daily frequency and severity of moderate to severe vasomotor symptoms

SECONDARY OUTCOMES:
vulvar and vaginal atrophy

REFERENCES:
- [Result] Hedrick RE. Low-dose estradiol gel 0.1% for the treatment of vasomotor symptoms associated with menopause. Expert Review of Obstetrics & Gynecology, 3(2): Pages 155-162, Mar 2008.